CLINICAL TRIAL: NCT04470349
Title: Comparison of Dynamic Distraction Systems in Proximal Interphalangeal Joint Fractures
Acronym: DYNAFIX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Waldfriede Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.1
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Proximal Interphalangeal Joint Fracture of the Hand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LITOS: Patients who received a LITOS dynamic distraction system after 31.12.2017
  Interventions: Device: LITOS
- Ligamentotaxor: Patients who received a Ligamentotaxor dynamic distraction system after 31.12.2017
  Interventions: Device: Ligamentotaxor

INTERVENTIONS:
Device: LITOS — Patients who received a LITOS dynamic distraction system after 31.12.2017
  Groups: LITOS
Device: Ligamentotaxor — Patients who received a Ligamentotaxor dynamic distraction system after 31.12.2017
  Groups: Ligamentotaxor

SUMMARY:
Fractures of the proximal interphalangeal joints continue to pose significant management challenges. Thus the aim of our study is to compare two dynamic finger joint distractors (Litos® and Ligamentotaxor®) in respect to the radiological standard follow-up examination and functional assessments.

ELIGIBILITY:
Inclusion Criteria:

* proximal interphalangeal fracture treated with external dynamic fixator
* Operative care <21 days from trauma
* Age between 18 and 90 years.
* Male and female

Exclusion Criteria:

- additional fractures or disabilities of the hand

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have sustained a proximal interphalangeal fracture treated with external dynamic fixator
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Disabilities of Arm, Shoulder and Hand (DASH) score | 3 months after explantation
  Disabilities as measured by the DASH scale; No Difficulty (1), Mild Difficulty (2), Moderate Difficulty (3), Severe Difficulty (4), Unable (5)

SECONDARY OUTCOMES:
Visual analogue scale (VAS) pain | 3 months after explantation
  From 0mm (no pain) to 100mm (maximum pain imaginable)
Functional assessment: Goniometry | 3 months after explantation
  ROM of each joint of the injured fingert with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Bock, MD, Principal Investigator — Waldfriede Hospital; Martin Lautenbach, MD, Study Chair — Waldfriede Hospital
Locations (1):
- Waldfriede Hospital, Berlin, Germany